CLINICAL TRIAL: NCT04096547
Title: A Prospective, Non-interventional, Multicenter Observational Study to Evaluate the Effectiveness and Safety of Rivaroxaban in Elderly NVAF Patients With or Without Renal Impairment
Brief Title: Rivaroxaban in Elderly NVAF Patients With or Without Renal Impairment
Acronym: XAIENT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Young Keun On, Professor, Samsung Medical Center
Other Study IDs: IRB 2019-06-078
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation; Rivaroxaban; Elderly; Renal Insufficiency
MeSH Terms: conditions — Atrial Fibrillation; Renal Insufficiency | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rivaroxaban — rivaroxaban for stroke prevention of atrial fibrillation

SUMMARY:
Study Type and Design Prospective, Observational Study Rivaroxaban in Elderly AF patients with or without renal impairment in Korea

This study will investigate effectiveness and safety in elderly patients, the result from well-designed and high-quality prospective clinical registry collected through real-world clinical practice is expected to resolve current medical unmet needs of rivaroxaban in Korean elderly patients.

Primary Study Objective(s) To investigate the effectiveness of rivaroxaban in elderly patients with NVAF, with or without renal impairment in Korea real-world clinical practice settings Secondary Study Objective(s) To see safety outcome including major bleeding, clinically non-major bleeding, all-cause mortality rivaroxaban in subgroup based on risk factor(eg. Renal impairment) physicians' treatment pattern in rivaroxaban

DETAILED DESCRIPTION:
Study Population Elderly patients with age ≥ 65 years with treatment naïve or treatment-experienced patients who are diagnosed with NVAF Expected number of patient enrollment is about 1200 patients, Samsung Medical Center is aim to enroll about 200 patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients with consent given
2. Elderly patients with age 65 ≥ years old
3. NVAF patients first time prescription to rivaroxaban or patients who started rivaroxaban treatment within 3 months

Exclusion Criteria:

1. Refusal to participate in this study or to give an informed consent
2. Patients with moderate to severe mitral stenosis
3. Patients with mechanical valve
4. Contraindication from rivaroxaban Korea SmPC

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with age ≥ 65 years with treatment naïve or treatment-experienced patients who are diagnosed with NVAF Expected number of patient enrollment is about 1200 patients,
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Composite incidence of stroke/ non-CNS SE | 1 year
  incidence of stroke/ non-CNS SE

SECONDARY OUTCOMES:
Bleeding incidence | 1 year
  Bleeding incidence

OTHER OUTCOMES:
renal function | 1 year
  CCl

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JY, Kim J, Park SJ, Park KM, Kim JS, Kim SH, Shim J, Choi EK, Kim DH, Oh IY, On YK; XAIENT Study Group. Comparison of High- and Low-Dose Rivaroxaban Regimens in Elderly East Asian Patients With Atrial Fibrillation. J Korean Med Sci. 2024 Mar 4;39(8):e72. doi: 10.3346/jkms.2024.39.e72. PMID 38442717